CLINICAL TRIAL: NCT03871894
Title: Metabolic and Clinical Effects of Enteral Nutrition Therapy: Measured Versus Estimated Energy and Substrate Requirements in Critically Ill Cirrhotics-A Randomized Controlled Trial
Brief Title: Indirect Calorimeter Based Study in Patients With Liver Cirrhosis
Acronym: METALIC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institute of Liver and Biliary Sciences, India (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ILBS-METALIC01
Record Dates: First submitted 2019-02-26; First posted 2019-03-12 (Actual); Last update posted 2022-10-24 (Actual); Status verified 2022-09

CONDITIONS: Liver Cirrhoses
Keywords: Indirect calorimeter; Resting energy expenditure; substrate utilization; nitrogen balance
MeSH Terms: interventions — Intensive Care Units

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control arm (Active Comparator): This is the group of critically ill cirrhotic patients on mechanical ventilator support who would receive the nutritional therapy as per the standard enteral nutritional practice in a critical care setting in cirrhotics till the period admitted in ICU(Intensive care unit) 35-40 Kcal/Kg IBW/day; 1.5g protein per kg per day.
  Interventions: Other: Indirect calorimetry based nutritional intervention till patient in ICU(Intensive care unit); Other: Standard and fixed nutritional intervention till patient in ICU
- Intervention arm (Experimental): This is the group of critically ill cirrhotic patients on mechanical ventilator support who would receive the nutritional therapy based on indirect calorimetry measurements till the period admitted in ICU(Intensive care unit); 1.5g protein per kg per day.
  Interventions: Other: Indirect calorimetry based nutritional intervention till patient in ICU(Intensive care unit); Other: Standard and fixed nutritional intervention till patient in ICU

INTERVENTIONS:
Other: Indirect calorimetry based nutritional intervention till patient in ICU(Intensive care unit) — Nutrition therapy based on measured energy expenditure by indirect calorimetry (IC) done alternate day till patient on ventilatory support and protein intake 1.5 g/kg IBW/day
Other: Standard and fixed nutritional intervention till patient in ICU — Fixed standard nutritional therapy 35-40 Kcal/Kg IBW/day and 1.5 g protein /Kg IBW/Day till patient on ventilator

SUMMARY:
Part I- Observational study In the first part , investigator would investigate and compare the energy requirements and substrate utilization in healthy subjects and in patients with liver cirrhosis of various etiologies across the disease severity state viz compensated, stable decompensated, critically ill cirrhotics. The investigator would also enroll patients with chronic kidney disease, critically ill patients of acute liver failure or acute on chronic liver failure as disease controls.

Part II- Randomized Controlled Study All the eligible, critically ill cirrhotic patients on mechanical ventilator support would be randomized to a control group (receiving the nutritional therapy as per the standard enteral nutritional practice in a critical care setting) or the intervention group (receiving enteral nutrition based on proposed measured requirements by Indirect calorimetry (IC) given till the patient is in ICU(Intensive care unit). The IC would be done thrice a week in both groups.

ELIGIBILITY:
Inclusion Criteria:

Disease groups:

• Patients with liver cirrhosis (diagnosis established based on routine clinical, biochemical and at least radiological, endoscopic or histological parameters.) admitted in Liver coma Intensive care unit and those admitted in ward.

Disease controls:

* Patients with Acute liver failure (diagnosis established based on routine clinical, biochemical and at least radiological parameters) admitted in Liver coma Intensive care unit
* Patients with severe acute pancreatitis (diagnosis established based on routine clinical, biochemical and at least radiological parameters) admitted in Liver coma Intensive care unit

Healthy Controls:

* Healthy subjects- Relatives of patients with no known chronic diseases (Chronic obstructive pulmonary disease, Coronary artery disease, Type 2 diabetes, Hypertension, Hypothyroidism, Koch's disease) or not on any long term medications.
* Patients with liver cirrhosis (diagnosis established based on routine clinical, biochemical and at least radiological, endoscopic or histological parameters.) admitted in Liver coma Intensive care unit who require mechanical ventilation

Exclusion Criteria:

* Age<18 years
* Active upper gastrointestinal bleeding
* If there are conditions which precluded IC, such as an FiO2 >60 %, failure to cooperate, agitation, seizure activity, spasticity, or positive end-expiratory pressure (PEEP) >10 mmHg.
* Pregnant women
* Refused to consent/ inability to obtain informed consent.
* Known long standing diabetic
* If there is any evidence of medical/surgical instability
* Hepatocellular carcinoma Extrahepatic malignancies
* With persistent gastrointestinal dysfunction and ileus
* Patients who would be readmitted to the ICU
* Known long standing diabetic
* Terminally ill patients on high inotropic support
* Acute liver failure
* If there is any evidence of medical/surgical instability
* If patients are taking any portion of nutrition by mouth.
* Pregnant women
* Refused to consent/ inability to obtain informed consent.
* Patient on CRRT- continuous renal replacement therapy
* Severe co morbidities such as Chronic kidney disease requiring maintenance dialysis, COPD and Cardiac pathologies (Acute myocardial infarction, heart failure, ).
* Hepatocellular carcinoma Extrahepatic malignancies
* Moribund patient with likely survival <24 hours
* Patients enrolled in other drug trials.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2019-03-12 (Actual); Primary Completion 2022-08-31 (Actual); Study Completion 2022-08-31 (Actual)

PRIMARY OUTCOMES:
Part 1: An Observational study | One day (Observational)
  Study groups :
  1. Healthy controls
  2. Disease Groups
     * Patients with liver cirrhosis (compensated and decompensated)
     * Critically ill cirrhotics on mechanical ventilator support
     * patients with chronic kidney disease (CKD) (stable,non dialyzed, non oliguric outpatients)
     * Critically ill patients with Acute liver failure (ALF) on mechanical ventilator support
     * Critically ill patients with Acute on chronic liver failure(ACLF) on mechanical ventilator support
     * Severe acute pancreatitis on mechanical ventilator support
  Comparison of the prevalence of hyper and hypo metabolism in patients with chronic liver disease(CLD) and healthy controls and other disease groups.
Part 2: A Randomized controlled trial | From date of enrollment until the date of ICU discharge /Leaving against medical advice, date of death from any cause, or off ventilatory support whichever comes first, assessed up to 28 days.
  Study group:Critically ill Cirrhotic: Diagnosed cases of liver cirrhosis with 2 or more organ failures (liver + renal/circulatory or respiratory failures) requiring ICU admission and on mechanical ventilator support meeting inclusion and exclusion criteria The difference in the duration of mechanical ventilation in critically ill ventilated patients with liver cirrhosis when the nutritional therapy delivered as per estimated energy requirements versus measured requirements

SECONDARY OUTCOMES:
Change in metabolic profile | The metabolic parameters would be assessed at the baseline, Day 7 and at Day 15 of enrollment
  The effect of nutritional therapy as per estimated energy requirements versus measured requirements in critically ill ventilated patients with liver cirrhosis on the Insulin resistance, ketone bodies, Non-esterified fatty acids (NEFA), amino acids profile and blood sugar levels would be studied
Change in inflammatory milieu | The inflammatory markers would be assessed at the baseline, Day 7 and at Day 15 of enrollment
  The effect of nutritional therapy as per estimated energy requirements versus measured requirements in critically ill ventilated patients with liver cirrhosis on the levels of interleukin 6 (IL-6), Tumor necrosis factor(TNF alfa), CRP(C reactive protein)would be studied
Change in clinical parameters | The clinical parameters would be assessed daily from the date of enrollment until the date of ICU discharge, date of death from any cause, or out of mechanical ventilatory support whichever comes first, assessed up to 28 days.
  The effect of nutritional therapy as per estimated energy requirements versus measured requirements in critically ill ventilated patients with liver cirrhosis ondevelopment of new onset infection, resolution of sepsis, renal function and length of stay in the ICU/hospital would be studied
Change in ventilatory and arterial blood gas parameters | The ventilatory and arterial blood gas parameters would be assessed daily from the date of enrollment until the date of ICU discharge, date of death from any cause, or out of mechanical ventilatory support whichever comes first, assessed up to 28 days.
  The effect of nutritional therapy as per estimated energy requirements versus measured requirements in critically ill ventilated patients with liver cirrhosis on ventilator parameters (FiO2, PEEP, PF ratio) and arterial blood gas parameters( PO2, PCO2, lactate, SpO2) would be studied
Change in nutritional parameters | The nutritional parameters would be assesses at regular intervals maximum upto 28 days
  The effect of nutritional therapy as per estimated energy requirements versus measured requirements in critically ill ventilated patients with liver cirrhosis on nutritional parameters( NUTRIC score, feed intolerance and would be studied
The association between energy metabolism, nutritional status and disease severity in patients with CLD | one day (Observational)
  The association between energy metabolism (resting energy expenditure- REE, substrate utilization and macronutrient oxidation), nutritional status (by body composition and anthropometry)and disease severity in patients with CLD (CTP and MELD scores) would be studied

CONTACTS AND LOCATIONS:
Overall Officials: Jaya Benjamin, Msc,PhD, Study Director — Institute of Liver and Biliary Sciences, sector D-1, Vasantkunj, New Delhi
Locations (1):
- ILBS, New Delhi, National Capital Territory of Delhi, India